CLINICAL TRIAL: NCT01811121
Title: Randomized, Prospective, Multicenter Blinding Singles With Arm A and Arm B Innovative Strategy Strategy Conventional
Brief Title: MEDICO-ECONOMIC EVALUATION OF SURGERY GUIDED BY FLUORESCENCE FOR THE OPTIMIZATION OF RESECTION OF GLIOBLASTOMAS
Acronym: RESECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-697
Record Dates: First submitted 2013-02-21; First posted 2013-03-14 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; 5ALA; fluorescence; resection
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-aminolévulinique acid (5-ALA) (Experimental): 5-aminolévulinique acid :microsurgical resection guided by fluorescence (CGF) in addition to the usual techniques of neuronavigation, after oral administration of 20mg/kg of 5-ALA 3-5 hours prior to surgical incision
  Interventions: Drug: 5-aminolévulinique acid (5-ALA)
- Placebo (Placebo Comparator): Laroscorbine :microsurgical excision guided solely by neuronavigation, after oral administration of a placebo 3 to 5 hours before the surgical incision
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-aminolévulinique acid (5-ALA) — oral administration of 20mg/kg of 5-ALA 3-5 hours before the surgical incision
  Other Names: Bras A
  Arms: 5-aminolévulinique acid (5-ALA)
Drug: Placebo — Oral administration of 1g of ascorbic acid LAROSCORBINE in 50ml of water 3 hours before surgery
  Other Names: Bras B
  Arms: Placebo

SUMMARY:
Glioblastoma is the most frequent primary malignant brain tumor in adults (3,000 new cases per year) and is characterized by a poor prognosis (median survival 12 months). Treatment is based mainly on surgical excision as complete as possible followed by an additional radiochemotherapy. The prognosis depends mainly on the quality of resection when it is macroscopically complete. Different techniques to support the surgical resection have been developed over the past 20 years. The reference technique is currently the intraoperative neuronavigation for guiding excision by matching the intraoperative tumor boundaries with those of the preoperative MRI. Its main drawback is the loss of precision during the resection related to changes in anatomical limits of the tumor.

The per-operative fluorescence-guided surgery (FGS) is an innovative alternative technique to support the surgical resection. The 5-aminolevulinic acid (5-ALA), a molecule absorbed by the patient before surgery is captured specifically by the tumor cells and transformed into a fluorochrome revealed intraoperatively by a light source length adapted wave with a set of lenses included in the microscope. Resection is thus guided by this fluorescence whose disappearance translates complete tumor resection.

Its interest is twofold:

* Increase the percentage of complete tumor resection.
* Improve disease-free survival and overall survival. The objective of the study is to compare the FGS to the intraoperative neuronavigation for the resection of glioblastoma, on a medical and economical level through a randomized, prospective, multicenter trial.

The annual number of patients likely to benefit of this technique in France is estimated at 2200 new cases.

DETAILED DESCRIPTION:
Main Outcome Measure: Percentage of patients with surgical resection of the tumor is complete, objectified by the absence of residual tumor on MRI early postoperative (within 48 hours) by a central committee of independent reading with qualitative analysis taking a contrast replay console for diagnostic use

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years with no upper age limit
* Competent adult patient.
* Patient affiliated to the National Health Insurance.
* Patient with an intra-cerebral supra-tentorial hemispheric, newly diagnosed and previously untreated, which MRI characteristics are suggestive of a glioblastoma.
* Indication for surgical treatment by excision.
* Brain tumor location distant from critical functional areas allowing a wide resection of contrast enhancement on imaging, the a priori character completely resectable has been validated by an evaluation committee composed of three surgeons
* No-cons contain medical surgery, ASA score below 4.
* Patient eligible for further treatment by radiotherapy and concurrent chemotherapy followed by adjuvant chemotherapy according to the so called Stupp scheme (standard protocol of adjuvant chemoradiotherapy)
* Negative pregnancy test for women of childbearing age.

Exclusion Criteria:

* Contraindications to performing an MRI (pacemaker).

  * Glioblastoma known and previously treated with surgery, radiotherapy and / or chemotherapy.
  * History of cancer.
  * Anatomical Location of the tumor-cons indicating a wide excision, neurosurgeon at the discretion of medical officer participating center.
  * Location tumor in the brain stem, the middle line, the basal ganglia and the posterior cranial fossa.
  * Patient with cons-indication to the achievement of further treatment with radiotherapy and concurrent chemotherapy followed by adjuvant chemotherapy according to the scheme proposed by Stupp. (1)
  * Patients with porphyria, renal insufficiency (creatinine> 177 μmolL), liver insufficency(gamma glutamyl transpeptidase> 100 U / L, prothrombin time <60%, bilirubin> 51μmol / L).
  * Patient refused to sign an informed consent form.
  * Ongoing participation of the patient to another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Comparison of complete tumor resection between the 2 arms | 48 hours
  Evidenced of complete resection (absence of residual tumor on early postoperative MRI (within 48 hours)) will be assessed by a central independent committee with qualitative analysis of contrast enhancement replay on a console for diagnostic use.

SECONDARY OUTCOMES:
Comparison of complete tumor resection between the 2 arms | less than 48 hours after surgery
  Evidenced of complete resection (absence of residual tumor on early postoperative MRI (within 48 hours)) will be assessed by the neurosurgeon who conducted the surgery and the neuro-radiologist who conducted the RMI with qualitative analysis of contrast enhancement replay during the initial clinical analysis

OTHER OUTCOMES:
Diagnostic value of the two intraoperative techniques | 60 months
  Evaluate the sensitivity, specificity, positive predictive value and negative by correlating the results of pathological analysis of resection edge with intraoperative findings of the surgeon at the end of resection.
Quantification of residual tumor (contrast enhancement) on MRI post-opératre early (before 48 hours) | before 48 hours
  It will be performed by three study investigators (Dr. Pallud, Department of Neurosurgery, Centre Hospitalier Sainte-Anne, Paris; Dr. Guyotat, D department of Neurosurgery, Hospices Civils de Lyon, Lyon, Dr. Metellus, neurosurgery department, Assistance Publique - Hôpitaux de Marseille) and read separately. The volume analysis will be done by segmentation using the OsiriX software on postoperative MRI and MRI pre-operative
Progression Free survival rate at 6 months | 6 months
  Progression is defined by the appearance of a new tumor lesion which minimum volume will be set to 0.175 cm3, by the increase of the residual tumor volume of 25% or more, or by the need to increase corticosteroid therapy. The period of progression free survival is defined as the time from the date of tumor resection and date of diagnosis of tumor progression or the date last news or date of endpoint. Progression Free survival rate at 6 months will be analyzed according to surgical approach used, according to the completeness or incompleteness of resection and by centers
Overall survival at 24 months | 24 months
  It will be estimated from the number of patients who died of whatever cause. The overall survival time is defined as the time between the date of tumor resection and date of death from any cause or date of last news or the date of endpoint. The overall survival at 24 months will be analyzed according to surgical approach used, according to the completeness or incompleteness of resection and by centers.
Overall survival at 60 months | 60 months
  It will be estimated from the number of patients who died of whatever cause. The overall survival time is defined as the time between the date of tumor resection and date of death from any cause or date of last news or the date of endpoint. The overall survival at 60 months will be analyzed according to surgical approach used, according to the completeness or incompleteness of resection and by centers.
Evaluation of Quality of life | every 3 months
  Evaluation of quality of life every 3 months using the EORTC questionnaire QLQ-C30 with the specific brain tumors module BN20.
Evaluation of early and late morbidity | in 8 days and late morbidity at 3 months
  Evaluation of early morbidity in 8 days and late morbidity at 3 months (neurological deficit, surgical site infection, secondary epilepsy, Karnofsky score, performance status WHO).
Comparison of surgical procedure duration between the 2 arms | 60 months
Medico-economic evaluation of the 2 procedure | 60 months
  Comparison of the differential cost effectiveness ratio between the 2 strategies

CONTACTS AND LOCATIONS:
Overall Officials: Jacques GUYOTAT, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Guyotat, Lyon, France

REFERENCES:
- [Result] Rioufol G, Derimay F, Roubille F, Perret T, Motreff P, Angoulvant D, Cottin Y, Meunier L, Cetran L, Cayla G, Harbaoui B, Wiedemann JY, Van Belle E, Pouillot C, Noirclerc N, Morelle JF, Soto FX, Caussin C, Bertrand B, Lefevre T, Dupouy P, Lesault PF, Albert F, Barthelemy O, Koning R, Leborgne L, Barnay P, Chapon P, Armero S, Lafont A, Piot C, Amaz C, Vaz B, Benyahya L, Varillon Y, Ovize M, Mewton N, Finet G; FUTURE Trial Investigators. Fractional Flow Reserve to Guide Treatment of Patients With Multivessel Coronary Artery Disease. J Am Coll Cardiol. 2021 Nov 9;78(19):1875-1885. doi: 10.1016/j.jacc.2021.08.061. PMID 34736563
- [Derived] Picart T, Pallud J, Berthiller J, Dumot C, Berhouma M, Ducray F, Armoiry X, Margier J, Guerre P, Varlet P, Meyronet D, Metellus P, Guyotat J; Members of RESECT study group:. Use of 5-ALA fluorescence-guided surgery versus white-light conventional microsurgery for the resection of newly diagnosed glioblastomas (RESECT study): a French multicenter randomized phase III study. J Neurosurg. 2023 Oct 13;140(4):987-1000. doi: 10.3171/2023.7.JNS231170. Print 2024 Apr 1. PMID 37856381